CLINICAL TRIAL: NCT05484388
Title: A Randomized Crossover Study to Evaluate Urine Leakage of Pant Type Absorbing Incontinence Products of Two Absorption Levels in a Home Care Environment
Brief Title: Evaluation of Urine Leakage of New Absorbing Incontinence Products in a Home Care Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Collaborators: Smerud Medical Research Germany Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SPRING
Record Dates: First submitted 2022-06-15; First posted 2022-08-02 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized pre-market feasibility clinical investigation designed to evaluate the clinical performance and safety of the investigational product in its intended target population.
  The clinical investigation is designed according to the ISO 14155:2020 as follows:
  Prospective.
  Randomized cross-over.
  Interventional but non-invasive.
  Decentralized in a home-care environment.
  A pairwise comparative study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SN2 (Experimental): new absorbing hygiene product with absorption level Normal.
  Interventions: Device: SN2
- SP3 (Experimental): new absorbing hygiene product with absorption level Plus.
  Interventions: Device: SP3
- TENA Proskin Pants Normal (Other): Reference product currently used by the participant (control for SN2).
  Interventions: Device: SN2
- TENA Pants Original Plus (Other): Reference product currently used by the participant (control for SP3).
  Interventions: Device: SP3

INTERVENTIONS:
Device: SN2 — Investigational device absorption level Normal
  Arms: SN2; TENA Proskin Pants Normal
Device: SP3 — Investigational device absorption level Plus
  Arms: SP3; TENA Pants Original Plus

SUMMARY:
The aim of this interventional but non-invasive, clinical investigation is to demonstrate the performance and safety of two new class I medical device Absorbing Hygiene Products developed by Essity.

The primary objective is to demonstrate for each of the new products that they provide protection to leakages similar to their corresponding standard of care devices already used on the market. The target population for this clinical investigation are community living individuals suffering from moderate to severe incontinence, who may receive care by a care giving relative, by one or more caregivers and are current users of TENA Pants of the respective absorption level.

DETAILED DESCRIPTION:
The clinical investigation will be conducted to demonstrate the performance and safety of two new class I medical device Absorbing Hygiene Products developed by Essity. The performance of the new design will be compared to that of the currently marketed TENA Pants, deemed state of the art.

To ensure that the personal preference of the study subjects are met, only current users of the marketed TENA pants will be recruited. To meet the objectives, the investigation is designed to be prospective, randomized, cross-over and interventional but not invasive with two different groups each testing one investigational-reference device pair matched to the currently used product at the time of inclusion. The study subjects will act as their own control, using one device for 10 (+ max. 3) days and then switching to the other device for additional 10 (+ max. 3) days. As for most users the avoidance of urinary leakages is the primary concern, this will be the primary outcome of the clinical investigation for each of the device pairs tested.

The used products will be collected, weighed and photographed. A subject/caregiver questionnaire will collect data on subject satisfaction and preferences. A skin health assessment will also be performed to evaluate any change in subject skin health before, during and at the end of the study.

Since the devices perform well in their intended use, leakage rate of each individual device is low, so a large number of devices needs to be tested per absorption level in order to obtain a robust assessment. Since the underlying incontinence condition is not affected by participation in the investigation, a sequential measurement series should be sufficient to meet the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* criteria to be eligible for this clinical investigation:

  1. Subject is diagnosed with moderate to severe urinary incontinence managed only with TENA Pants absorbent hygiene products of size Medium or Large with the same absorption level that is used in the study since at least 4 weeks.
  2. Subject is living at home and should have a care giving relative supported by a professional caregiver giver to manage daily activities and incontinence related tasks.
  3. Subject is willing and able to provide informed consent and to participate in the clinical investigation or has a legally designated representative willing to provide informed consent on behalf of the subject.
  4. Care giving relative is willing and able to provide informed consent to participate in the clinical investigation.
  5. If incontinence is managed by pharmaceuticals, the dose regime is stable.
  6. Subject and care giving relative (if any) are over 18 years of age.
  7. Post-menopausal women or no longer of child-bearing potential

Exclusion Criteria:

1. Subject is cared for in a professional establishment or is institutionalized.
2. Subject has severe incontinence product related skin problems corresponding to scores equal to or higher than 4 in the skin health assessment, as judged by the investigator.
3. Subject suffers from regular faecal incontinence more than once a week.
4. Subject has any type of urinary catheter(s) resulting in improved/treated urinary incontinence.
5. Any other condition that may make participation in the clinical investigation inappropriate, as judged by investigator.
6. Subject or care giving relative is incapable or unwilling to collect used products and fill out the bag label required for the clinical investigation.
7. Participation in another investigational study of a drug, biologic, or medical device within 30 days prior to entering the clinical investigation or planned during the clinical investigation as well as prior participation in this investigation
8. Subject is pregnant or nursing or of childbearing potential.
9. Investigator suspects that subject or care giving relative has an alcohol or drug addiction.
10. Subject and/or caregiving relative is closely affiliated with or in hierarchical dependency of the Sponsor, PI, or CRO involved in this study
11. Subject's incontinence is currently managed by more than 1 type of AHP's
12. Surgery or hospitalization less than 4 weeks prior to study inclusion or planned surgery hospitalization during study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Reported number of urinary leakages | 20 days
  The proportion of products experiencing urine leakage over the 10 day test period is compared between the investigational and reference product. Labels are used to collect this information for each used product

SECONDARY OUTCOMES:
Incidence of safety events | 20 days
  The number and severity of reported safety events are collected and compared for the intervention and reference products
Product Satisfaction questionnaire | 20 days
  To evaluate caregiver perception of and experience in using the products. Overall satisfaction score with investigational product as compared to the reference product using a 5-point likert scale.
Skin health questionnaire | 20 days
  To evaluate subject's skin health for the investigational product as compared to the reference product as part of the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kilian Pankert, MD, Principal Investigator — Diakonissen-Stiftungs-Krankenhaus Speyer
Locations (1):
- Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer, Germany

IPD SHARING:
Plan to Share IPD: No